CLINICAL TRIAL: NCT02749903
Title: A Phase II Study of Enzalutamide (NSC# 766085) for Patients With Androgen Receptor Positive Salivary Cancers
Brief Title: Enzalutamide for Patients With Androgen Receptor Positive Salivary Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A091404; NCI-2015-01706 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Salivary Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide (Other): Patients receive 160 mg enzalutamide orally once daily (1 cycle=28 days). Patients will remain on therapy until progression of disease or development of unacceptable toxicities or patient or physician withdrawal. Patients will undergo radiographic imaging every 2 months while on study treatment in order to determine response.
  Interventions: Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — oral

SUMMARY:
This study will test any good and bad effects of the study drug called enzalutamide. Enzalutamide could shrink the cancer but it could also cause side effects. Researchers hope to learn if the study drug will shrink the cancer by at least 30% compared to its present size, in at least 1 out of 5 patients. Enzalutamide is not FDA approved to treat salivary gland cancer, but it has already been FDA-approved to treat other cancers.

DETAILED DESCRIPTION:
This single arm Phase II trial will assess the best overall response associated with enzalutamide in patients with AR-positive salivary cancers. Given that this will be one of the first prospective studies ever conducted for AR-positive salivary cancers, and there are currently no standard therapies known to be effective for this disease, the investigators will adopt a best overall response (BOR) of 5% as the null hypothesis and BOR of 20 % as the alternative hypothesis. In addition to response, this study will also evaluate the progression-free survival (PFS), overall survival (OS), adverse events, and will also try to identify molecular predictors of response by examining genomic and transcriptional elements of androgen receptor biology.

The primary and secondary objectives of the study:

Primary objective

To evaluate the rate of best overall response associated with enzalutamide in patients with AR-positive salivary cancers

Secondary objectives

1. To evaluate the progression-free survival (PFS) of AR-positive salivary cancer patients treated with enzalutamide
2. To evaluate the overall survival (OS) of AR-positive salivary cancer patients treated with enzalutamide
3. To evaluate the safety/tolerability of enzalutamide for patients with AR-positive salivary cancer

Patients are followed up to 3 years after study enrollment.

ELIGIBILITY:
1. Documentation of Disease - Histologic Documentation: Histologically proven diagnosis of salivary cancer by central pathology review. Receptor status: AR expression detected by immunohistochemistry by central review.
2. Disease status - Measurable disease as defined in the protocol. Locally advanced/unresectable (as determined by local surgeon) OR metastatic disease.
3. Prior Treatment

   * Any number of prior lines of therapy
   * No treatment with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, or radiation ≤ 28 days before study registration. No treatment with nitrosourea or mitomycin ≤ 42 days before study registration
   * No prior therapy with enzalutamide (previous chemotherapy and/or other AR-targeted approaches is allowed).
4. Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects. A female of childbearing potent is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (ie, has had menses at any time in the preceding 12 consecutive months). For women of childbearing potential only, a negative pregnancy test done ≤ 5 days prior to registration is required.
5. Age ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
7. No History of the following:

   * prior brain metastases
   * leptomeningeal disease
   * seizures
   * class 3 or 4 congestive heart failure
   * uncontrolled hypertension (systolic BP > 170 mmHg or diastolic BP > 105 mmHg)
   * major surgery ≤ 4 weeks of registration
8. Required Initial Laboratory Values:

   * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   * Platelet Count ≥ 100,000/mm3
   * Creatinine ≤ 1.5 x ULN Upper Limit of Normal (ULN) OR
   * Calculated Creatinine Clearance ≥ 30 mL/min
   * Total Bilirubin ≤ 1.5 x ULN
   * AST/ALT ≤ 3.0 x ULN
9. Concomitant medications- Chronic concomitant treatment with strong CYP2C8 inhibitors is not allowed. Patients must discontinue the drug ≥ 14 days prior to registration. Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug ≥ 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2028-07-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (287):
- United States (287):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute?Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Laurens, Clinton, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Inova Fairfax Hospital-Woodburn Infusion Clinic, Annandale, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Ho AL, Foster NR, Zoroufy AJ, Campbell JD, Worden F, Price K, Adkins D, Bowles DW, Kang H, Burtness B, Sherman E, Morton R, Morris LGT, Nadeem Z, Katabi N, Munster P, Schwartz GK. Phase II Study of Enzalutamide for Patients With Androgen Receptor-Positive Salivary Gland Cancers (Alliance A091404). J Clin Oncol. 2022 Dec 20;40(36):4240-4249. doi: 10.1200/JCO.22.00229. Epub 2022 Jul 22. PMID 35867947

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enzalutamide
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 4
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 25
    1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: The best overall response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients.
Time Frame: Up to 32 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Enzalutamide
Number analyzed (Participants) | 46
percentage of patients | 4.3 [0.5 to 14.8]

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 32 months post study enrollment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 46
months | 5.6 [3.7 to 7.5]

3. Secondary Outcome: Number of Patients Experiencing at Least One Grade 3+ Adverse Event Using CTCAE Version 4.0
Description: The number of patients experiencing at least one grade 3+ adverse event using CTCAE version 4.0 is summarized below.
Time Frame: 30 days post-treatment, up to 32 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 46
Participants | 22

ADVERSE EVENTS:
Time Frame: Up to 30 days post-treatment, up to 32 months
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 27/46
Serious Adverse Events (participants affected / at risk) | 15/46
Other Adverse Events (participants affected / at risk) | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=46)
Heart failure (Cardiac disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Bone infection (Infections and infestations) | 1 (3)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=46)
Anemia (Blood and lymphatic system disorders) | 11 (22)
Atrial fibrillation (Cardiac disorders) | 1 (4)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (12)
Heart failure (Cardiac disorders) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 2 (5)
Hearing impaired (Ear and labyrinth disorders) | 1 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (32)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (36)
Dry mouth (Gastrointestinal disorders) | 4 (22)
Dysphagia (Gastrointestinal disorders) | 3 (22)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (8)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (13)
Oral pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (3)
Toothache (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 5 (7)
Edema limbs (General disorders) | 2 (3)
Facial pain (General disorders) | 1 (4)
Fatigue (General disorders) | 40 (205)
Fever (General disorders) | 1 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (8)
Localized edema (General disorders) | 9 (22)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (3)
Pain (General disorders) | 6 (24)
Gum infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (4)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alkaline phosphatase increased (Investigations) | 5 (9)
Aspartate aminotransferase increased (Investigations) | 6 (14)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (2)
Investigations - Other, specify (Investigations) | 1 (20)
Lymphocyte count decreased (Investigations) | 8 (25)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 21 (44)
White blood cell decreased (Investigations) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 10 (37)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (26)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (5)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (12)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 13 (41)
Dysgeusia (Nervous system disorders) | 3 (24)
Dysphasia (Nervous system disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 2 (7)
Headache (Nervous system disorders) | 3 (11)
Paresthesia (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Seizure (Nervous system disorders) | 1 (4)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (7)
Depression (Psychiatric disorders) | 2 (6)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (30)
Libido decreased (Psychiatric disorders) | 1 (6)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 10 (72)
Gynecomastia (Reproductive system and breast disorders) | 8 (67)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (13)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (28)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 22 (123)
Hypertension (Vascular disorders) | 34 (207)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02749903/Prot_SAP_000.pdf